CLINICAL TRIAL: NCT03203564
Title: An Adaptive, Randomized, Double-blind, Single-center, Placebo-controlled Phase I Study Evaluating ECG Effects, Safety and Pharmacokinetics of Single Ascending Doses of [6R]-5,10-Methylene Tetrahydrofolate (Modufolin® for Injection, 100mg) in Healthy Male Volunteers
Brief Title: Study Evaluating ECG Effects, Safety, Tolerability and Pharmacokinetics of Single Doses of Modufolin (Arfolitixorin) in Healthy Volunteers Tetrahydrofolate in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: ISO-FF-001
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Phase I Study in Healthy Volunteers to Evaluate ECG Effect

STUDY DESIGN:
Intervention Model Description: An adaptive, randomized, double-blind, single-center, placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: IMP (Modufolin® for Injection, 100 mg) and Placebo are not identical in appearance and all efforts will be made at the clinic in order to maintain the blind. Both the IMP and the placebo will be masked in such a way that study subjects and study staff will remain blinded during the study. An un-blinded study nurse will prepare the IMP/placebo for injection and will administer the IMP/placebo to the study subject. The un-blinded study nurse performing the dose administration will not be involved in any study-specific assessments or evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modufolin® for injection, 200, 350 and 500 mg/m2 (Active Comparator): Three cohorts, 8 subjects will be randomised to Modufolin ® for injection 100 mg
  Interventions: Drug: Modufolin (arfolitixorin)
- 0.9% NaCl sterile solution (Placebo Comparator): Three cohorts, 3 subjects will be randomised to placebo
  Interventions: Drug: Modufolin (arfolitixorin)

INTERVENTIONS:
Drug: Modufolin (arfolitixorin) — Thirty-three eligible and consenting subjects will be included in 3 cohorts, 11 subjects in each cohort, Within each cohort, subjects will be randomized to receive either placebo (3 subjects) or Modufolin® for injection, 100mg (8 subjects)
  Other Names: arfolitixorin

SUMMARY:
The purpose of this study is to evaluating ECG effects, safety, tolerability and pharmacokinetics of single ascending dose of Modufolin® in healthy male volunteers

DETAILED DESCRIPTION:
An adaptive randomised, double-blind, single-centre, placebo-controlled Phase I study evaluating ECG effects, safety, tolerability and PK of single ascending doses of Modufolin® for Injection, 100 mg in healthy male volunteers. Thirty-three (33) eligible and consenting subjects will be included in 3 cohorts, 11 subjects in each cohort. Within each cohort, subjects will be randomised to receive either placebo (3 subjects) or Modufolin® for Injection, 100 mg (8 subjects). There will be 3 pre-defined ascending dose-levels. Additional dose levels may be considered if recommended by the internal Safety Review cCommittee. There will be an interval between each dose level to allow time for safety data to be analyzed and evaluated by the iSRC. The iSRC will have the choice to decide to escalate the dose as planned, reduce or increase the dose escalation step, repeat the dose, reduce the dose or terminate the study. The total study duration for the subjects will be approximately 5 weeks and there will be in total 3 visits to the clinic. Subjects will be screened for eligibility according to study-specific inclusion/exclusion criteria within 4 weeks prior to start of stud treatment (Visit 1; Screening visit). The subjects will be confined to the research clinic from the evening before dosing (Day -1) until 24 hrs post dose (Days 1 and 2). The subjects should be fasting overnight (8 hrs) before IMP/placebo administration until 4 hrs post-dose. A Follow-up Visit will be performed 5 to 10 days after dose administration of for each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide a written informed consent for participation in the study.
2. Healthy male subject aged 18-60 years inclusive.
3. Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 and weight at least 50 kg and no more than 100 kg at screening and body surface area ≤ 2 m2
4. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Willing to use condom and highly effective contraceptive methods with a failure rate of < 1% to prevent pregnancy1 and drug exposure to a partner and refrain from donating sperm from the date of dosing until 3 months after dosing of the IMP/placebo.

Exclusion Criteria:

* 1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or subject´s ability to participate in the study.

  2. Any clinically significant illness, medical/surgical procedure or trauma within four weeks of the first administration of IMP/placebo. 3. Any planned major surgery within the duration of the study. 4. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV). 5. After 10 minutes (min) supine rest at the time of screening, any vital signs values outside the following ranges:
  * Systolic BP > 150 mm Hg
  * Diastolic BP > 90 mm Hg
  * Pulse < 40 or > 85 beats per min 6. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.

    7. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to Modufolin® (i.e., folate derivatives). 8. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two weeks prior to the administration of IMP/placebo, except occasional intake of paracetamol (maximum 2000 mg/day; and not exceeding 3 000 mg/week), at the discretion of the Investigator and nasal decongestants without cortisone or antihistamine for a maximum of 10 days, at the discretion of the Investigator. 9. Regular use of any prescribed or non-prescribed medication which could influence folate and vitamin B12 status within 30 days prior to the administration of IMP/placebo.

    10. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment with less than three months between administration of last dose and first dose of IMP/placebo in this study. Subjects consented and screened but not dosed in previous phase I studies are not excluded. 11. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit. 12. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP/placebo. 13. Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse.

    14. Intake of xanthine and/or taurine containing energy drinks within two days prior to screening.

    15. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to dosing. 16. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a database of healthy volunteers at CTC and from advertising in media, including social media.
Pre-assignment Details: Subjects were screened for eligibility according to study-specific inclusion/exclusion criteria within four weeks prior to start of study treatment (Visit 1; Screening Visit).
Groups:
- 200 mg/m2 of Modufolin®: 8 subjects were treated with 200 mg/m2 of Modufolin® as an intravenous bolus injection.
- 350 mg/m2 of Modufolin®: 8 subjects were treated with 350 mg/m2 of Modufolin® as an intravenous bolus injection.
- 500 mg/m2 of Modufolin®: 8 subjects were treated with 500 mg/m2 of Modufolin® as an intravenous bolus injection.
- Placebo: 9 subjects were treated with placebo as an intravenous bolus injection.
Period: Overall Study
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Started | 8 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 9 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 9 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 8 | 7 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 8 | 8 | 8 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline QTcF (ΔQTcF)
Description: At each nominal time point specified in the CSP, up to 10 ECG replicates were extracted with TQT Plus methods. TQT Plus ECG extraction technique: Twelve-lead ECGs were extracted from continuous recordings (Holter recordings) prior to and serially after IMP administration at time points as shown in the Schedule of events. Subjects were supinely resting for at least 10 min prior to time points for ECG recordings.
  The 12-lead Holter and ECG equipment were supplied and supported by iCardiac Technologies, Inc.
  For all ECG parameters, baseline is defined as the average of the measured ECG intervals from the three pre-dose time points (45, 30, and 15 min pre-dose) on Day 1.
Time Frame: Pre-dose at following timepoints -2 h, -45 min, -30 min, -15 min. Then at following timepoints; 0, 5 min, 15 min, 30 min, 1 h, 2h, 3h, 4h, 5h, 6h, 8h, 12h and 24h post-dose.
Population: The QT/QTc Analysis Set includes all subjects in the Safety Analysis Set with measurements at baseline as well as on-treatment with at least one post-dose time point with a valid ΔQTcF (change from baseline QTcF) value.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
msec
  End of infusion | 2.8 (2.85) | 9.2 (2.84) | 8.5 (2.87) | 1.1 (2.69)
  5 min post-dose | 11.2 (2.28) | 9.1 (2.28) | 22.4 (2.31) | 0.0 (2.16)
  15 min post-dose | 3.1 (1.48) | 7.5 (1.47) | 12.4 (1.51) | 0.2 (1.40)
  30 min post-dose | 1.2 (1.43) | 2.5 (1.42) | 4.2 (1.47) | 0.8 (1.36)
  1 h post-dose | -1.2 (1.38) | -0.7 (1.38) | -0.9 (1.42) | 1.4 (1.32)
  2 h post-dose | -3.5 (1.97) | -1.7 (1.96) | 1.0 (1.99) | 0.7 (1.86)
  3 h post-dose | -2.8 (2.58) | -0.8 (2.58) | 0.9 (2.60) | 3.8 (2.44)
  4 h post-dose | -3.3 (2.70) | 0.7 (2.70) | 0.0 (2.72) | 2.6 (2.55)
  5 h post-dose: number analyzed (Participants) | 8 | 7 | 8 | 9
  5 h post-dose | 5.4 (3.25) | 2.6 (3.37) | 0.8 (3.27) | 11.5 (3.07)
  6 h post-dose | -0.8 (2.73) | -2.5 (2.72) | -6.7 (2.75) | 6.4 (2.58)
  8 h post-dose | -5.5 (2.91) | -5.5 (2.90) | -7.7 (2.93) | -0.9 (2.75)
  12 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  12 h post-dose | -4.5 (2.86) | -6.6 (2.86) | -4.1 (2.95) | 2.8 (2.70)
  24 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  24 h post-dose | -5.9 (2.85) | -8.1 (2.84) | -4.6 (3.01) | -1.3 (2.69)
Statistical Analysis 1: Comparison: 200 mg/m2 of Modufolin® vs 350 mg/m2 of Modufolin® vs 500 mg/m2 of Modufolin® vs Placebo; The primary analysis of QTcF was based on a linear mixed-effects model with change-from-baseline QTcF as the dependent variable, time (categorical), treatment, and time-by-treatment interaction as fixed effects, and baseline QTcF as a covariate. The least-squares (LS) mean and 2-sided 90 % CIs have been calculated for the contrast "Modufolin® versus placebo" at each dose of Modufolin® and each post-dose time point; Test type: Other; Mean Difference (Final Values) = 7.4, 90% CI 2-sided [0.68 to 14.12] — Parameter estimate is done for Placebo-corrected change-from baseline QTcF (ΔΔQTcF) for Modufolin 500 mg/m2 at end of infusion

2. Secondary Outcome: Relationship Between ΔΔQTc and Modufolin® (and Metabolites) Plasma Concentrations
Description: Predicted ΔΔQTcF interval at geometric mean Cmax for 5,10-MTHF, THF, and 5-Formyl-THF and geometric mean concentration of 5-Methyl-THF observed at 5 minutes post-dose The relationship between plasma concentrations of 5,10-MTHF, THF, 5-Methyl-THF, and 5-Formyl-THF, and change-from-baseline QTcF (ΔQTcF) was quantified using a linear mixed-effects modeling approach with separate analyses for each of the analytes (5,10-MTHF, THF 5-Methyl-THF, and 5-Formyl-THF) initially, with ΔQTcF as the dependent variable, plasma concentration of 5,10-MTHF (or THF, 5-Methyl-THF, or 5-Formyl-THF) as a continuous covariate (i.e., 0 for placebo), centered baseline QTcF as an additional covariate, treatment (active = 1 or placebo = 0) and time (i.e., time point) as categorical factors, and a random intercept and slope per subject. The degrees of freedom estimates were determined by the Kenward-Roger method.
Time Frame: 5 minute post-dose time point
Measure: Geometric Mean (90% Confidence Interval); unit: msec / ng/mL
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin®
Number analyzed (Participants) | 8 | 8 | 8
msec / ng/mL
  5,10-MTHF | 24111.78 [19194.04 to 30289.52] | 51566.94 [46351.78 to 57368.87] | 69012.28 [60609.82 to 78579.59]
  THF | 15995.29 [13750.28 to 18606.83] | 29386.77 [26812.58 to 32208.09] | 44018.37 [40400.31 to 47960.44]
  5-Methyl-THF | 218.18 [176.04 to 270.40] | 544.01 [435.70 to 679.25] | 333.09 [279.56 to 396.86]
  5-Formyl-THF | 296.43 [114.76 to 765.71] | 567.17 [414.42 to 776.22] | 379.33 [333.23 to 431.81]
  ΔΔQTcF | 4.15 [0.97 to 7.33] | 13.25 [9.36 to 17.14] | 19.88 [15.40 to 24.35]

3. Secondary Outcome: Change-from-baseline Heart Rate (ΔHR)
Description: The analysis was based on the change-from-baseline post-dosing values. The same (by-time point analysis) model was used as described for QTcF. For all ECG parameters, baseline is defined as the average of the measured ECG intervals from the three pre-dose time points (45, 30, and 15 min predose) on Day 1.
Time Frame: as for outcome 1
Population: QT/QTc population.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
bpm
  End of infusion | 2.6 (1.91) | 2.7 (1.91) | 2.0 (1.92) | -2.1 (1.80)
  5 min post-dose | 8.2 (2.56) | 7.4 (2.55) | 13.3 (2.56) | 0.0 (2.41)
  15 min post-dose | 3.9 (1.63) | 3.6 (1.63) | 2.6 (1.64) | -1.6 (1.53)
  30 min post-dose | 3.3 (2.00) | 1.3 (2.00) | 3.0 (2.00) | -0.7 (1.88)
  1 h post-dose | 5.0 (1.90) | 0.0 (1.90) | -0.9 (1.91) | -1.3 (1.79)
  2 h post-dose | 3.2 (1.52) | -0.1 (1.52) | -2.6 (1.53) | -1.8 (1.43)
  3 h post-dose | 2.2 (1.47) | 0.3 (1.46) | 0.3 (1.47) | -2.3 (1.38)
  4 h post-dose | 1.7 (1.82) | 2.0 (1.82) | 0.2 (1.83) | -3.3 (1.72)
  5 h post-dose: number analyzed (Participants) | 8 | 7 | 8 | 9
  5 h post-dose | 11.9 (2.06) | 12.4 (2.12) | 8.9 (2.06) | 9.5 (1.94)
  6 h post-dose | 8.3 (2.52) | 12.5 (2.52) | 6.2 (2.53) | 5.4 (2.38)
  8 h post-dose | 8.1 (2.24) | 8.0 (2.23) | 2.5 (2.24) | 2.1 (2.11)
  12 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  12 h post-dose | 7.6 (2.41) | 5.3 (2.41) | 3.6 (2.54) | 0.6 (2.27)
  24 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  24 h post-dose | 6.0 (2.80) | 5.7 (2.80) | 8.0 (3.00) | 8.6 (2.64)

4. Secondary Outcome: Change-from-baseline PR (ΔPR)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: QT/QTc population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
msec
  End of infusion | -1.6 (2.08) | -4.4 (2.08) | -2.1 (2.08) | -1.6 (1.96)
  5 min post-dose | -1.5 (2.07) | -4.5 (2.07) | -3.1 (2.07) | -0.1 (1.96)
  15 min post-dose | -2.3 (2.61) | -1.2 (2.61) | 0.2 (2.61) | 3.8 (2.46)
  30 min post-dose | -1.7 (2.11) | -3.7 (2.11) | 1.3 (2.11) | 2.9 (1.99)
  1 h post-dose | -5.2 (1.89) | -3.6 (1.89) | -0.3 (1.89) | 0.4 (1.79)
  2 h post-dose | -4.1 (2.13) | -4.1 (2.13) | 1.1 (2.13) | 3.1 (2.01)
  3 h post-dose | -5.3 (2.14) | -4.2 (2.14) | -1.6 (2.14) | 1.2 (2.02)
  4 h post-dose | -5.2 (1.84) | -4.6 (1.84) | -2.1 (1.84) | 1.4 (1.74)
  5 h post-dose: number analyzed (Participants) | 8 | 7 | 8 | 9
  5 h post-dose | -8.8 (2.59) | -7.1 (2.71) | -7.8 (2.59) | -3.5 (2.44)
  6 h post-dose | -9.4 (2.04) | -8.4 (2.04) | -5.8 (2.04) | -3.9 (1.93)
  8 h post-dose | -8.6 (2.62) | -7.2 (2.62) | -4.3 (2.62) | -5.6 (2.47)
  12 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  12 h post-dose | -7.9 (3.12) | -1.5 (3.12) | -6.9 (3.22) | -1.7 (2.94)
  24 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  24 h post-dose | -5.9 (2.77) | -5.6 (2.77) | -6.4 (2.88) | -6.8 (2.61)

5. Secondary Outcome: Change-from-baseline QRS (ΔQRS)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: QT/QTc population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
msec
  End of infusion | -0.1 (0.27) | -0.2 (0.27) | -0.1 (0.27) | 0.5 (0.25)
  5 min post-dose | -0.7 (0.28) | -0.8 (0.28) | -1.2 (0.28) | 0.0 (0.26)
  15 min post-dose | -0.2 (0.25) | -0.3 (0.25) | -0.1 (0.25) | 0.0 (0.24)
  30 min post-dose | -0.7 (0.27) | 0.0 (0.27) | -0.5 (0.27) | 0.0 (0.26)
  1 h post-dose | -0.2 (0.26) | 0.1 (0.26) | 0.2 (0.26) | 0.0 (0.24)
  2 h post-dose | -0.2 (0.22) | 0.0 (0.22) | -0.1 (0.22) | -0.1 (0.21)
  3 h post-dose | 0.0 (0.30) | -0.1 (0.31) | -0.4 (0.30) | 0.2 (0.29)
  4 h post-dose | 0.1 (0.39) | -0.5 (0.39) | 0.2 (0.38) | 0.9 (0.36)
  5 h post-dose: number analyzed (Participants) | 8 | 7 | 8 | 9
  5 h post-dose | 0.4 (0.47) | 0.4 (0.49) | 0.1 (0.47) | 0.2 (0.45)
  6 h post-dose | -0.3 (0.52) | -0.4 (0.52) | -0.8 (0.52) | -0.7 (0.49)
  8 h post-dose | -0.3 (0.53) | -0.3 (0.53) | -0.5 (0.53) | -0.6 (0.50)
  12 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  12 h post-dose | 0.5 (0.56) | 0.3 (0.56) | -0.6 (0.58) | -1.0 (0.53)
  24 h post-dose: number analyzed (Participants) | 8 | 8 | 7 | 9
  24 h post-dose | 0.0 (0.45) | 0.4 (0.45) | -0.9 (0.47) | -0.9 (0.42)

6. Secondary Outcome: Number of Participants With Categorical QTcF Outliers
Description: QTcF outliers per absolute category across treatment groups and QTcF outliers per change-from-baseline category (ΔQTcF)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Participants
  No. participants with QTcF > 450 and ≤ 480 msec | 0 | 0 | 1 | 0
  No. participants with QTcF > 480 and ≤ 500 msec | 0 | 0 | 0 | 0
  No. participants with QTcF > 500 msec | 0 | 0 | 0 | 0
  No. participants with ΔQTcF of > 30 and ≤ 60 msec | 0 | 0 | 2 | 0
  No. participants with ΔQTcF > 60 msec | 0 | 0 | 0 | 0

7. Secondary Outcome: Categorical Outliers for HR, PR Interval, QRS Interval
Description: Categorical Analysis of outliers for HR, PR, and QRS intervals
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Participants
  HR changes >25% decrease from baseline to <50 bpm | 0 | 0 | 0 | 0
  HR changes >25% increase from baseline to >100bpm | 0 | 0 | 0 | 0
  PR changes > 25% increase from baseline to >200ms | 0 | 0 | 0 | 0
  QRS changes > 25% increase from baseline to >120ms | 0 | 0 | 0 | 0

8. Secondary Outcome: Categorical Analysis for T Wave Morphology
Description: Categorical T-wave morphology analysis and measurement of PR and QRS intervals were fully performed manually in three of the 10 ECG replicates at each time point. Final quality control and diagnostic interpretations were performed by the study cardiologist. When the results for each time point were compiled in the final data set, the comparison was made between ECG parameters from the three manually reviewed ECGs versus the 10 ECG replicates for quality control purposes. No treatment emergent T wave morphology changes were observed. In addition to the T-wave categorical analysis, the presence of abnormal U-waves was noted.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Participants
  Flat | 0 | 0 | 0 | 0
  Notched (+) | 0 | 0 | 0 | 0
  Biphasic | 0 | 0 | 0 | 0
  Normal (-) | 0 | 0 | 0 | 0
  Notched (-) | 0 | 0 | 0 | 0
  U wave presence | 0 | 0 | 0 | 0

9. Secondary Outcome: Physical Examination
Description: A complete physical examination included assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities.
  Physical examination findings were categorized as Normal, Abnormal non-clinical significant (NCS), and Abnormal clinical significant (CS).
Time Frame: At visit 1 (screening) and follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Participants
  Abnormal NCS - Visit 1 | 0 | 0 | 1 | 0
  Abnormal CS - Visit 1 | 0 | 0 | 0 | 0
  Abnormal NCS - Follow-up | 0 | 0 | 0 | 0
  Abnormal CS - Follow-up | 0 | 0 | 0 | 0

10. Secondary Outcome: Systolic Blood Pressure
Description: Systolic and diastolic BP and pulse were measured in supine position after 10 min of rest.
Time Frame: Predose at following timepoints: At screening (visit 1) and at -15 min (visit 2). Postdose at following timepoints: 3h, 5h, 8 h and 24h (visit 2) and at visit 3 (follow-up visit).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
mmHg
  Screening | 115.50 (7.60) | 121.25 (7.07) | 116.63 (9.56) | 125.56 (14.82)
  Visit 2 Day 1 (-00:15) | 111.38 (10.94) | 109.38 (9.36) | 117.38 (8.11) | 123.67 (24.63)
  Visit 2 Day 1 (03:00) | 108.88 (7.12) | 105.00 (6.89) | 112.50 (9.29) | 111.22 (7.87)
  Visit 2 Day 1 (05:00) | 115.50 (5.61) | 115.00 (8.50) | 120.88 (7.94) | 113.00 (13.32)
  Visit 2 Day 1 (08:00) | 118.50 (9.06) | 113.88 (6.75) | 115.63 (5.83) | 114.89 (10.61)
  Visit 2 Day 2 | 117.75 (9.29) | 114.13 (5.77) | 120.88 (8.46) | 119.00 (10.02)
  Follow-up | 121.38 (8.93) | 115.63 (11.03) | 119.38 (10.21) | 122.11 (12.24)

11. Secondary Outcome: Diastolic Blood Pressure
Description: Systolic and diastolic BP and pulse were measured in supine position after 10 min of rest.
  There were no clinically relevant mean changes over time or any individual changes assessed as clinically significant with regards to any of the vital signs parameters.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
mmHg
  Screening | 68.63 (5.21) | 69.75 (8.51) | 72.25 (8.01) | 73.56 (11.75)
  Visit 2 Day 1 (-00:15) | 69.63 (3.74) | 65.88 (6.42) | 75.38 (2.77) | 69.56 (9.06)
  Visit 2 Day 1 (03:00) | 69.00 (6.89) | 64.38 (7.37) | 72.63 (5.71) | 65.56 (11.20)
  Visit 2 Day 1 (05:00) | 65.63 (5.88) | 62.38 (5.04) | 72.25 (7.15) | 67.00 (11.16)
  Visit 2 Day 1 (08:00) | 69.00 (7.29) | 64.50 (3.89) | 70.25 (6.36) | 66.22 (9.59)
  Visit 2 Day 2 | 71.50 (10.23) | 69.38 (4.50) | 74.25 (5.47) | 71.11 (8.15)
  Follow-up | 68.25 (4.53) | 70.25 (7.81) | 71.00 (8.07) | 70.11 (7.99)

12. Secondary Outcome: Vital Signs: Pulse
Description: as for outcome 11
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
bpm
  Screening | 59.50 (5.21) | 66.50 (9.38) | 62.00 (11.24) | 63.22 (12.88)
  Visit 2 Day 1 (-00:15) | 55.25 (5.44) | 52.00 (8.60) | 56.38 (5.58) | 54.44 (11.34)
  Visit 2 Day 1 03:00) | 56.25 (5.50) | 53.13 (11.01) | 53.75 (4.95) | 50.33 (6.60)
  Visit 2 Day 1 (05:00) | 65.38 (4.00) | 65.25 (9.66) | 66.00 (11.60) | 61.44 (8.92)
  Visit 2 Day 1 (08:00) | 60.25 (6.82) | 59.00 (5.83) | 56.75 (7.21) | 55.67 (7.23)
  Visit 2 Day 2 | 59.38 (9.53) | 57.63 (8.91) | 61.75 (13.48) | 61.22 (11.31)
  Follow-up | 66.25 (9.04) | 67.88 (12.91) | 69.25 (16.26) | 67.44 (14.47)

13. Secondary Outcome: Safety Laboratory Measurements
Description: The following safety laboratory parameters were assessed:
  Clinical Chemistry: Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Albumin, Aspartate aminotransferase (AST), Bilirubin (total and conjugated), Calcium, Chloride, Creatinine, Magnesium, Phosphorous, Potassium, Sodium, Urea nitrogen, Uric acid. Haematology: Haematocrit, Haemoglobin (Hb), Platelet count, Red blood cell (RBC) count, White blood cell (WBC) count with differential count. Urinalysis (dip stick):Glucose, Erythrocytes, Nitrite, Protein, Specific gravity, pH.
Time Frame: Pre-dose at screening (visit 1) and -2h (visit 2). Post-dose at following timepoints: 24 h (visit 2) and at follow-up (visit 3)
Measure: Number; unit: Clinically relevant changes
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Clinically relevant changes | 0 | 0 | 0 | 0

14. Secondary Outcome: Frequency, Seriousness and Intensity of AEs
Description: An overall summary of AEs occurring after first administration of IMP (TEAE) is presented by treatment
Time Frame: From start of IMP administration to follow-up visit
Population: FAS
Measure: Number; unit: Adverse events
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Adverse events
  No. of TEAEs | 8 | 8 | 16 | 2
  No. of subject-unique TEAEs | 8 | 7 | 16 | 2
  Subject-unique related TEAEs | 7 | 4 | 14 | 0
  SAEs | 0 | 0 | 0 | 0

15. Secondary Outcome: Plasma PK Characteristics: C0
Description: The mean back-extrapolated concentration at time 0 h (C0) was calculated for MTHF
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h. pre-dose to 24 h post-dose
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 0
ng/mL | 34200 (10300) | 78300 (12600) | 99000 (23100) |

16. Secondary Outcome: Plasma PK Characteristics: C5min
Description: Measured concentration at 5 min post dose (C5min) of MTHF and 5-Formyl-THF
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
ng/mL
  MTHF | 24600 (6480) | 52200 (8530) | 70100 (13100) |
  5-Formyl-THF | 443 (432) | 609 (240) | 374 (83.2) |

17. Secondary Outcome: Plasma PK Characteristics: AUClast
Description: Pharmacokinetic parameters were calculated for test item MTHF, and for the following metabolites: 5-Formyl-THF, 5-Methyl-THF, and THF, if data permitted
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
h*ng/mL
  MTHF | 10900 (1680) | 19700 (1990) | 31100 (3210) |
  THF | 31800 (3780) | 53100 (10000) | 90100 (17500) |
  5-Methyl-THF | 23400 (4470) | 38500 (6380) | 47400 (7540) |

18. Secondary Outcome: Plasma PK Characteristics: AUClast/Dose
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: (h*ng/mL)/mg
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
(h*ng/mL)/mg
  MTHF | 29.2 (5.27) | 29.8 (2.74) | 32.9 (4.93) |
  THF | 85.0 (11.8) | 80.1 (14.0) | 95.0 (19.2) |
  5-Methyl-THF | 62.7 (12.5) | 58.3 (9.87) | 49.9 (7.91) |
  5-Formyl-THF | 2.33 (1.97) | 1.24 (1.22) | 0.343 (0.580) |

19. Secondary Outcome: Plasma PK Characteristics: Timepoint for Last Measured Plasma Concentration (Tlast)
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification (LLOQ).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
hour
  MTHF | 4.38 (1.95) | 5.37 (1.30) | 6.75 (2.31) |
  THF | 7.01 (1.52) | 8.01 (0.0178) | 8.75 (2.12) |
  5-Methyl-THF | 24.0 (0.0339) | 24.0 (0.0980) | 23.8 (0.135) |
  5-Formyl-THF | 3.41 (2.94) | 3.00 (2.92) | 1.40 (2.67) |

20. Secondary Outcome: Plasma PK Characteristics: t1/2
Description: Pharmacokinetic parameters were calculated for test item MTHF, and for the following metabolites: 5-Formyl-THF, 5-Methyl-THF, and THF, if data permitted:
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
hour
  MTHF: number analyzed (Participants) | 3 | 4 | 5 | 0
  MTHF | 0.989 (0.936) | 1.87 (0.634) | 2.03 (0.780) |
  THF | 1.35 (0.211) | 1.51 (0.267) | 1.59 (0.370) |
  5-Methyl-THF | 5.54 (0.714) | 5.66 (0.644) | 5.84 (0.634) |

21. Secondary Outcome: Plasma PK Characteristics: CL
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
L/h
  MTHF: number analyzed (Participants) | 3 | 4 | 5 | 0
  MTHF | 38.6 (1.84) | 35.5 (3.05) | 30.6 (5.14) |
  THF | 11.6 (1.47) | 12.6 (2.58) | 10.7 (2.37) |
  5-Methyl-THF | 15.6 (3.11) | 16.5 (2.63) | 19.1 (3.49) |

22. Secondary Outcome: Plasma PK Characteristics: Vss
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: litre
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
litre
  MTHF: number analyzed (Participants) | 3 | 4 | 5 | 0
  MTHF | 18.1 (9.38) | 20.4 (6.10) | 18.5 (6.07) |
  THF | 21.8 (3.30) | 24.9 (4.17) | 21.6 (4.43) |
  5-Methyl-THF | 138 (28.4) | 153 (27.4) | 181 (27.9) |

23. Secondary Outcome: Plasma PK Characteristics: Cmax
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
ng/mL
  THF | 16400 (3610) | 29600 (3970) | 44400 (6090) |
  5-Methyl-THF | 2490 (450) | 3950 (755) | 4740 (484) |
  5-Formyl-THF: number analyzed (Participants) | 3 | 8 | 8 | 0
  5-Formyl-THF | 642 (474) | 619 (257) | 386 (75.3) |

24. Secondary Outcome: Plasma PK Characteristics: Tmax
Description: as for outcome 17
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h.
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
hour
  THF | 0.267 (0.334) | 0.123 (0.0786) | 0.300 (0.179) |
  5-Methyl-THF | 3.12 (0.835) | 3.50 (1.07) | 3.63 (0.519) |
  5-Formyl-THF: number analyzed (Participants) | 3 | 8 | 8 | 0
  5-Formyl-THF | 0.0778 (0.0255) | 0.102 (0.0601) | 0.142 (0.145) |

25. Secondary Outcome: Plasma PK Characteristics: Cmax/Dose for Metabolite 5-Formyl-THF
Description: Pharmacokinetic parameters were calculated for test item MTHF, and for the following metabolites: 5-Formyl-THF, 5-Methyl-THF, and THF, if data permitted. Only the metabolite 5-Formyl-THF has values above LLOQ and are presented below.
Time Frame: Pre-dose at -15 min and post-dose at following timepoints: 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h
Population: All samples analysed from the subjects given placebo were below Lower Limit of Quantification.
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 0
ng/mL/mg | 1.73 (1.33) | 0.934 (0.379) | 0.407 (0.0826) |

26. Secondary Outcome: Number of Subjects With AEs
Description: An overall summary of subjects with AEs occurring after first administration of IMP (TEAE), number of related TEAEs and number of withdrawals due to TEAEs are presented by treatment
Time Frame: From start of IMP administration to follow-up visit
Population: FAS
Measure: Number; unit: Subjects
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Subjects
  Subjects with at least one TEAE | 6 | 5 | 8 | 1
  Subjects with at least one related TEAE | 5 | 3 | 8 | 0
  Withdrawals due to TEAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from start of IMP administration to last subject last visit, thus during a period of little less than 2 months.
Arm/Group | 200 mg/m2 of Modufolin® | 350 mg/m2 of Modufolin® | 500 mg/m2 of Modufolin® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 6/8 | 5/8 | 8/8 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg/m2 of Modufolin® (N=8) | 350 mg/m2 of Modufolin® (N=8) | 500 mg/m2 of Modufolin® (N=8) | Placebo (N=9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia oral (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Non-disclosure agreement that prohibits the PI to communicate results without a prior permission from the sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03203564/SAP_000.pdf
  • Study Protocol (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT03203564/Prot_001.pdf